CLINICAL TRIAL: NCT04148014
Title: Emotion Regulation Group Skills Training: A Pilot Study of an add-on Treatment for Eating Disorders in a Clinical Setting
Brief Title: Emotion Regulation Group Skills Training for Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Maria Zetterqvist, Prinicipal investigator, Region Östergötland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/472-32
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Eating Disorders; Emotions; Skill, Coping
Keywords: eating disorders; young adults; emotion regulation skills
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: A pilot study without randomization or controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjunctive Emotion Regulation Skills Training (Experimental): Participants will receive a 5 session once a week group emotion regulation skills training adjacent to treatment as usual provided by the eating disorder unit at the child and adolescent psychiatric clinic, Linköping, Sweden.
  Interventions: Behavioral: An Adjunctive Emotion Regulation Skills Training

INTERVENTIONS:
Behavioral: An Adjunctive Emotion Regulation Skills Training — The adjunctive emotion regulation skills training is delivered in a group format once a week during 5 weeks to young adults with eating disorders together with treatment as usual

SUMMARY:
Emotion regulation difficulties appear to play a role in the development and maintenance of several eating disorders. This pilot study aims at examining whether a short add-on group skills training in emotion regulation for young adults with different eating disorders is feasible in a psychiatric clinical setting. We also investigate if the treatment increases knowledge of emotions, and decreases self-reported difficulties with emotion regulation, alexithymia, symptoms of eating disorder, anxiety and depression, as well as clinical impairment.

Six skills training groups were piloted with a total of 29 participants (M = 21.41 years, SD = 1.92). The treatment consists of five sessions dealing with psychoeducation about emotions and emotion regulation skills training. Paired samples t-test was used to compare differences between before-and-after measures.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled as a patient at the eating disorder unit at eh child- and adolescent psychiatric clinic in Linköping, Sweden
* Having an eating disorder diagnosis as primary diagnosis.
* Being between the ages of 18-25 years
* Having sufficient knowledge of the Swedish language

Exclusion Criteria:

* Clinical diagnosis of schizophrenia
* Clinical diagnosis of psychosis
* Clinical diagnosis of severe autism spectrum disorder
* Having a cognitive disability
* Having ongoing drug or alcohol abuse
* Clinical diagnosis of bipolar disorder
* Insufficient knowledge of the Swedish language

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on biological sex.
Enrollment: 39 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Difficulties with Emotion Regulation Scale (DERS) | Change from baseline at 5 weeks
  Difficulties with Emotion Regulation Scale measures difficulties with emotion regulation. It contains a total of 36 items that are rated on a Likert scale between 1-5. Total score ranges between 36-180 with higher scores indicating more difficulties with emotion regulation. The scale has 6 subscales: nonacceptance (ranging from 6-30); goals (ranging from 5-25); impulse (ranging from 6-30); awareness (ranging from 6-30); strategies (ranging from 8-40) and clarity (ranging from 5-25).
Toronto Alexithymia Scale (TAS-20) | Change from baseline at 5 weeks
  Toronto Alexithymia Scale measures alexithymia. It contains a total of 20 items with 3 subscales (difficulties describing feelings: 7 items ranging from 7-35, difficulties identifying feelings: 5 items ranging from 5-25 and externally oriented thinking: 8 items ranging from 8-40). Total scores range from 20-100 with higher scores indicating higher levels of alexithymia.
Eating Disorder Examination Questionnaire (EDE-Q). | Change from baseline at 5 weeks
  The Eating Disorder Examination Questionnaire (EDE-Q) is the self-report version of Eating Disorder Examination (EDE) and measures the characteristics of eating disorders. The 6.0 version used in this study consists of 28 items. EDE-Q is scored on a 7-point Likert scale, from "no days" to "every day" and higher scores indicate higher eating pathology. The total score ranges from 0-196. The questionnaire comprises a total scale and subscales for restraint, eating concerns, shape concerns and weight concerns.
The Clinical Impairment Assessment Questionnaire (CIA) | Change from baseline at 5 weeks
  The Clinical Impairment Assessment Questionnaire (CIA) measures the psychosocial impairment of eating disorders. It focuses on the last 28 days and consists of 16 items, graded on a Likert scale from "Not at all" to "A lot". Higher scores indicate higher level of secondary psychosocial impairment and the total scores ranges from 0-48. The CIA is designed to be completed immediately after filling in a measure of current eating disorder features that covers the same time frame (e.g., the EDE-Q).

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale, self-report version (MADRS-S). | Change from baseline at 5 weeks
  Montgomery Åsberg Depression Rating Scale measures symptoms of depression. Its main purpose is to monitor the development of symptoms during treatment. The scale consists of 9 items, which are graded from zero to six. Total scores range from 0-54. Higher scores indicate higher level of depression symptoms.
Beck's Anxiety Inventory (BAI) | Change from baseline at 5 weeks
  Beck's Anxiety Inventory measures symptoms of anxiety with 21 items rated on a four-graded scale (0-3). Total scores range from 0-63. Higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Zetterqvist, PhD, Principal Investigator — Region Östergötland
Locations (1):
- Region Ostergotland BUP-kliniken, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmqvist Larsson K, Lowen A, Hellerstedt L, Bergcrona L, Salerud M, Zetterqvist M. Emotion regulation group skills training: a pilot study of an add-on treatment for eating disorders in a clinical setting. J Eat Disord. 2020 Apr 3;8:12. doi: 10.1186/s40337-020-00289-1. eCollection 2020. PMID 32266070